CLINICAL TRIAL: NCT02639871
Title: Validation of Molecular Neuroimaging Biomarkers in Huntington's Disease in View of Therapeutic Trials Targeting the Krebs Cycle
Brief Title: Dynamic Neuroimaging Biomarkers in Huntington's Disease
Acronym: HDeNERGY
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CEA (Unknown)
Responsible Party: Sponsor
Other Study IDs: P140708; 2015-A00793-46 (Other: IDCRB)
Record Dates: First submitted 2015-12-15; First posted 2015-12-28 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Brain Neuroimaging Biomarkers in Huntington Disease
Keywords: Huntington disease; Neuroimaging metabolic biomarker
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- healthy volunteers: 31P-MR Spectroscopy and CEST for Validation of MRI/MRS methods
- HD presymptomatic individuals: General medical exam Clinical assessment with illness rating scales: Unified Huntington's Disease Rating Scale Total Motor Score (UHDRS) and Total Functional Capacity (TFC), 31P-MR Spectroscopy and CEST
- early affected HD patients: General medical exam Clinical assessment with illness rating scales: UHDRS and TFC, 31P-MR Spectroscopy and CEST
- Controls: General medical exam Clinical assessment with illness rating scales: UHDRS and TFC, 31P-MR Spectroscopy and CEST

SUMMARY:
There is no curative treatment available today in Huntington disease (HD) despite the identification of the mutated gene 20 years ago. Nonetheless, safe and promising therapeutic strategies targeting brain energy metabolism are now becoming available.

In view of the small effect sizes of any clinical parameter in HD, robust neuroimaging biomarkers reflecting brain energy metabolism are therefore urgently needed to better assess the potential of therapeutics targeting the mitochondria, and especially the Krebs cycle. Identifying such biomarkers at the presymptomatic phase in HD also provides a unique window for therapeutic intervention, which can be used as a proof-of-concept for the real challenge of tomorrow's medicine: the prevention of neurodegeneration HDeNERGY is an observational study consisting of the transfer of methods from preclinical to clinical studies and their application in HD. HDeNERGY aim at optimizing MRI/MRS methods to study the dynamics of brain energy metabolism. At the CENIR (Centre de neuro-imagerie et de recherche, Paris) the determination of creatine kinase rate will be first validated in healthy volunteers (n=20) and then applied to the selected cohort of early affected HD patients (n=20), presymptomatic individuals (n=20) and controls (n=20) together with the methods previously validated in HD patients (Mochel et al., 2012b) to determine the ratio of inorganic phosphate (Pi)/ phosphocreatine (PCr) during visual stimulation in presymptomatic individuals. The Chemical Exchange Saturation Transfer (CEST) method on the 3T clinical scanner of CENIR will be first validated in healthy volunteers (n=20) and then applied to the selected cohort of early affected HD patients (n=20), presymptomatic individuals (n=20) and controls (n=20).

The cerebral synthesis rate of creatine phosphate and of brain glutamate concentrations and pH values will be compared between controls, HD patients and HD presymptomatic individuals, and correlated with clinical parameters (age, BMI, UHDRS).

DETAILED DESCRIPTION:
Compelling evidence indicate a key role of energy defects in neurodegenerative diseases (NDs). These defects would constitute extremely informative functional biomarkers of disease states and progression. Such functional biomarkers could be used as readouts for therapeutic efficacy in clinical trials, especially for drugs targeting brain energy metabolism. Magnetic Resonance Imaging (MRI) and Magnetic Resonance Spectroscopy (MRS) are likely the most promising approaches to validate brain biomarkers linked to energy metabolism. However, existing methods allowing "static" measures of metabolites concentrations offer only a fragmented vision of brain energy metabolism in NDs. The validation of novel and "dynamic" methods is urgently needed. Our project addresses this challenge for Huntington disease (HD).

Our study is an observational study consisting of the transfer of methods from preclinical to clinical studies and their application in HD.

This study comprises two period:

* Period 1: transfer of 31P saturation transfer and CEST methods from preclinical to clinical MRS/MRI platforms and the validation of these methods in healthy individuals;
* Period 2: compare brain metabolic markers in early individuals affected by HD, presymptomatic individuals and controls, using 31P saturation transfer and CEST methods.

The primary objectives are:

Using 31P saturation transfer and CEST methods, the primary objective is to compare novel metabolic biomarkers between controls and HD carriers (patients and presymptomatic individuals).

Assessment criterion:

Comparison between controls, HD patients and HD presymptomatic individuals of the cerebral synthesis rate of creatine phosphate and of brain glutamate concentrations and pH values

The secondary objectives are:

* To develop/optimize 31P MRS/CEST methods to study the dynamics of brain energy metabolism in humans
* To improve the understanding and "modeling" the nature of energy deficits in HD
* To look for correlations between brain energy profiles and clinical scores.

Assessment criteria:

* Validation of the 31P MRS and CEST methods in healthy volunteers.
* Combination and integration of the 31P MRS and CEST data in order to obtain a model of energy deficits in HD.
* Correlations between creatine phosphate synthetic rate and clinical parameters (age, BMI, UHDRS); correlations between glutamate concentrations and clinical parameters; correlations between pH values and clinical parameters.

Ancillary studies:

The investigators wish to compare brain energy parameters (creatine phosphate synthetic rate, glutamate concentrations, pH values) with systemic metabolic markers (profiles of plasma metabolites obtained from metabolomic and lipidomic studies).

ELIGIBILITY:
Inclusion criteria

Healthy Volunteers Period 1:

* At least 18 years of age
* Signature of the informed consent
* Covered by social security

Participants Period 2:

* At least 18 years of age
* Signature of the informed consent
* Covered by social security
* Presymptomatic individuals: Positive genetic test with CAG repeat length > 39 in HTT gene, UHDRS score < 5
* Early affected patients: Positive genetic test with CAG repeat length > 39 in HTT gene and UHDRS score between 5 and 40
* BMI between 18 and 30

Non-inclusion criteria

Healthy Volunteers Period 1:

* Contra-indications to MRI (claustrophobia, metallic or material implants)
* History of severe head injury
* Participation in another trial
* Pregnancy and breastfeeding
* Inability to understand information about the protocol
* Persons deprived of their liberty by judicial or administrative decision
* Adult subject under legal protection or unable to consent.
* Unwillingness to be informed in case of abnormal MRI

Participants Period 2:

* Contra-indications to MRI (claustrophobia, metallic or material implants)
* Additional psychiatric or neurological conditions / Additional major comorbidities
* History of severe head injury
* Participation in another trial
* Pregnancy and breastfeeding
* Inability to understand information about the protocol
* Persons deprived of their liberty by judicial or administrative decision
* Adult subject under legal protection or unable to consent.
* Unwillingness to be informed in case of abnormal MRI
* Treatment with tetrabenazine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Period 1: healthy volunteers; Period 2: presymptomatic individuals, early affected HD patients and controls
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Cerebral synthesis rate of creatine phosphate | 1 day
  Comparison between controls, HD patients and HD presymptomatic individuals of the cerebral synthesis rate of creatine phosphate
Cerebral brain glutamate concentrations | 1 day
  Comparison between controls, HD patients and HD presymptomatic individuals of brain glutamate concentrations
Cerebral pH values. | 1 day
  Comparison between controls, HD patients and HD presymptomatic individuals of pH values

SECONDARY OUTCOMES:
Measure concentration of brain phosphocreatine (PCr) and glutamate using 31P MRS and gluCEST respectively in healthy volunteers | 1 day
  The 31P MRS will allow to measure the synthesis rate of PCr at different time points - rest, visual stimulation and recovery after stimulation. The rate of PCr synthesis will give an indication on the integrity of the rate of creatine-kinase.
  gluCEST will allow to measure the regional distribution of glutamate in the brain in order to create glutamate maps.
Data integration of rate of phosphocreatine (PCr) synthesis and gluatamate concentrations. | 1 day
  A model of energy deficit in HD can be created by looking at the correlation between the rate of PCr synthesis, glutamate maps and the disease.
Correlations between the ratio of phosphocreatine concentration at different time point and age of participants | 1 day
Correlations between the ratio of phosphocreatine concentration at different time points and BMI of participants. | 1 day
Correlations between creatine phosphate synthetic rate and UHDRS | 1 day
Correlations between glutamate concentrations and age | inclusion visit
Correlations between glutamate concentrations and BMI | inclusion visit
Correlations between glutamate concentrations and UHDRS | 1 day
Correlations between pH values and age | 1 day
Correlations between pH values and BMI | 1 day
Correlations between pH values and UHDRS | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Fanny MOCHEL, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- APHP - Pitié Salpetriere Hospital, Paris, France